CLINICAL TRIAL: NCT02248272
Title: The Effects of Meal Frequency on Glucose, Insulin, and Insulin Sensitivity in Women With Polycystic Ovary Syndrome (PCOS), People at High Risk for Developing Type 2 Diabetes and People With Type 2 Diabetes
Brief Title: Effect of Meal Frequency on Glycemic Control of People at High Risk or Diagnosed With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meropi Kontogianni (Other)
Collaborators: Agricultural University of Athens (Other); National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor-Investigator, Meropi Kontogianni, Assistant Professor, Harokopio University
Organization: Harokopio University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8062; HUA (Other: Harokopio University)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Impaired Glucose Tolerance; Hyperinsulinism; Poor Glycemic Control; Hyperglycemia; Insulin Sensitivity
Keywords: Polycystic ovary syndrome; Type 2 Diabetes; Hyperinsulinemia; Meal frequency
MeSH Terms: conditions — Glucose Intolerance; Hyperinsulinism; Hyperglycemia; Insulin Resistance; Polycystic Ovary Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Polycystic Ovary Syndrome (Experimental): 40 women with PCOS followed one of two isocaloric weight maintenance diets (isocaloric diet with 3 meals or isocaloric diet with 6 meals), tailored to individual energy needs, with the same macronutrient composition (40% carbohydrates, 25% protein, 35% fat). The energy and carbohydrate contribution for the 3 meals' diet was 20% at breakfast, 50% at lunch, 30% at dinner, whereas for the 6 meals' diet was 20% at breakfast, 10% at morning snack, 30% at lunch, 10% at afternoon snack, 20% at dinner, 10% at before bedtime snack. Each intervention lasted 12 weeks and there was no wash out period.
  Interventions: Other: Isocaloric diet with 3 meals; Other: Isocaloric diet with 6 meals
- Impaired Glucose Tolerance (Experimental): 35 individuals with Impaired Glucose Tolerance (IGT) followed one of two isocaloric weight maintenance diets (isocaloric diet with 3 meals or isocaloric diet with 6 meals), tailored to individual energy needs, with the same macronutrient composition (45% carbohydrates, 20% protein, 35% fat). The energy and carbohydrate contribution for the 3 meals' diet was 20% at breakfast, 50% at lunch, 30% at dinner, whereas for the 6 meals' diet was 20% at breakfast, 10% at morning snack, 30% at lunch, 10% at afternoon snack, 20% at dinner, 10% at before bedtime snack. Each intervention lasted 12 weeks and there was no wash out period.
  Interventions: Other: Isocaloric diet with 3 meals; Other: Isocaloric diet with 6 meals
- Type 2 Diabetes (Experimental): 12 individuals diagnosed with type 2 diabetes followed one of two isocaloric weight maintenance diets (isocaloric diet with 3 meals or isocaloric diet with 6 meals), tailored to individual energy needs, with the same macronutrient composition (45% carbohydrates, 20% protein, 35% fat). The energy and carbohydrate contribution for the 3 meals' diet was 20% at breakfast, 50% at lunch, 30% at dinner, whereas for the 6 meals' diet was 20% at breakfast, 10% at morning snack, 30% at lunch, 10% at afternoon snack, 20% at dinner, 10% at before bedtime snack. Each intervention lasted 12 weeks and there was no wash out period.
  Interventions: Other: Isocaloric diet with 3 meals; Other: Isocaloric diet with 6 meals

INTERVENTIONS:
Other: Isocaloric diet with 3 meals — Isocaloric diet with 3 meals in order to maintain volunteers' weight, tailored to individual energy needs, with the same macronutrient composition. The volunteers were free to choose the foods they used to consume before. However, in order to assist them to adapt to the different meal frequency, individualized instructions were given to all volunteers before their entry to the study. An example of a 7-day diet menu was prescribed for both diet programs and analytical food exchange lists of different food groups were also provided.
Other: Isocaloric diet with 6 meals — Isocaloric diet with 6 meals in order to maintain volunteers' weight, tailored to individual energy needs, with the same macronutrient composition. The volunteers were free to choose the foods they used to consume before. However, in order to assist them to adapt to the different meal frequency, individualized instructions were given to all volunteers before their entry to the study. An example of a 7-day diet menu was prescribed for both diet programs and analytical food exchange lists of different food groups were also provided.

SUMMARY:
This study investigated any potential associations between two isocaloric diets with different meal frequency (3 meals versus 6 meals) and glycemic control in people at high diabetes risk (lean and overweight/obese women with PCOS, individuals with hyperinsulinemia, individuals with impaired glucose tolerance) and diagnosed with diabetes.

DETAILED DESCRIPTION:
The effect of meal frequency on diabetes risk markers (e.g. glucose and insulin metabolism) has been studied in several studies so far, both in healthy individuals and in individuals being at risk for diabetes mellitus, with or without concurrent weight loss. In addition, few studies have investigated the effect of different meal frequency on glycemic control in patients with diabetes mellitus under conditions of weight maintenance. However, the results regarding the ideal number of meals remain controversial.

To our best knowledge, there is no study available that has investigated the effect of meal frequency on glucose and insulin metabolism in lean and obese women with PCOS, in lean and obese individuals with hyperinsulinemia and impaired glucose tolerance, and in obese individuals with type 2 diabetes, independently of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* The presence of type 2 diabetes was defined according to the current diagnostic criteria: (a) HbA1c ≥ 6.5%, (b) fasting plasma glucose ≥126 mg/dl (7.0 mmol/l). (c) 2-h plasma glucose ≥ 200 mg/dl (11.1 mmol/l) during an oral glucose tolerance test (OGTT), using a glucose load containing the equivalent of 75 g anhydrous glucose dissolved in water, or (d) a random plasma glucose ≥ 200 mg/dl (11.1 mmol/l) in patients with classic symptoms of hyperglycemia or hyperglycemic crisis.
* PCOS was defined according to the Rotterdam criteria (Rotterdam 2004) which include the presence of two or more of the following features: chronic oligoovulation or anovulation (fewer than six menstrual periods in the previous year), androgen excess (serum total testosterone >70 mg/dl) and polycystic ovaries.

Exclusion Criteria:

* Insulin sensitizers, i.e. metformin, contraceptives, steroids or any medications known to affect glucose, insulin or reproductive hormones for at least the last 6 months.
* Serious health problems like cardiovascular, liver or kidney diseases.
* Volunteers who were on diet, using medications affecting body mass or who had experienced a change in body weight ≥ 4.5 kg or a change in physical activity within the 6 months preceding the study onset were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Serum levels of glucose | 6 months
  Clinically useful change in serum glucose, defined as the restoration of glucose within normal limits during the 2-hour oral glucose tolerance test.

SECONDARY OUTCOMES:
Serum levels of insulin | 6 months
  Clinically useful change in serum insulin, defined as the restoration of insulin within normal limits during the 2-hour oral glucose tolerance test. Improved insulin sensitivity.
HbA1c | 6 months
  Clinically useful change in HbA1c.
Lipidemic profile | 6 months
  Normal serum levels of cholesterol, High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL) and Triglycerides.

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Study Director — Agricultural University of Athens; Meropi Kontogianni, PhD, Principal Investigator — Harokopio University of Athens